CLINICAL TRIAL: NCT02329275
Title: HPV as a Possible Cause of Azoospermia
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Consultant, Ph.D., Odense University Hospital
Other Study IDs: Lab.Reprod.Biol.- Odense.02
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: HPV in Testis Tissue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Azoospermic men
  Interventions: Procedure: Testicular biopsy
- Men with proven fertility
  Interventions: Procedure: Testicular biopsy

INTERVENTIONS:
Procedure: Testicular biopsy

SUMMARY:
Azoospermia is found in 5-20% of all men suffering from infertility, and in more than 20% azoospermia remains unexplained. The investigators suggest, that HPV may be an etiological factor in azoospermia and reduced sperm production.

The investigators plan to examine the occurrence of HPV in testicular tissue from 100 azoospermic men and to compare with the HPV occurrence in testicular tissue from a control group of 40 normal, healthy men undergoing vasectomy. Since HPV, in a recent Danish study, was detected on sperm in 16% of 188 randomly selected semen donors, the investigators also plan to examine the occurrence of HPV on sperm ejaculated during the last week before vasectomy. If HPV should be found in testicular tissue from men belonging to the control group, it will be highly relevant to compare with the HPV occurrence on sperm ejaculated from the men in concern.

A Linear Array HPV Genotyping Kit from Roche will be used for detection of HPV in testicular tissue and ejaculates. In total, with this test kit 37 HPV genotypes are examined for, including 13 high risk types.

ELIGIBILITY:
Inclusion Criteria:

* Men with azoospermia (Group 1) and proven fertile men undergoing vasectomy (Group 2)

Exclusion Criteria:

* Men with testicular abnormalities (Group 2)
* Men who do not understand the purpose and possible consequences of the study (both groups)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Unselected azoospermic men referred to the fertility clinic Group 2: Proven fertile men referred for vasectomy
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
HPV DNA in testicular tissue | Two years
  In tissue from both azoospermic and proven fertile men

SECONDARY OUTCOMES:
HPV DNA in ejaculates | Two years
  In ejaculates from the proven fertile men

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Odense University Hospital, Odense, Denmark